CLINICAL TRIAL: NCT04739358
Title: A Phase 1/2 Open-Label Study To Determine a Central Nervous System (CNS) Dose and Schedule Of Tepotinib Alone Or In Combination With Other Relevant Tyrosine Kinase Inhibitors (TKIs) In Adult Participants With MET-Driven NSCLC
Brief Title: CNS Dose Escalation/Expansion of Tepotinib in MET-driven NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to lack of lack of enrollment and difficult patient population.
Sponsor: Criterium, Inc. (Industry)
Collaborators: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01AT21-MET
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Advanced Non-Small Cell Lung Cancer With MET Mutations
Keywords: Non-Small Cell Lung Cancer, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tepotinib

STUDY DESIGN:
Intervention Model Description: Phase I - Two arms (Monotherapy and Combination therapy) with a primary endpoint of Dose Limiting Toxicity Phase II - Two arms Monotherapy Cohort: Primary endpoint is Intracranial Objective Response Rate; Combination Cohort: Primary endpoint is overall and extracranial ORR among patients treated with the combination of tepotinib and concurrent TKI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): * Dose Escalation Phase for participants with MET-driven NSCLC.
  * Dose Expansion Phase: CNS Efficacy Dose Expansion Cohort for participants with MET-driven NSCLC and measurable CNS disease.
  Interventions: Drug: Tepotinib
- Combination Therapy (Experimental): * Dose Escalation Phase for participants with evidence of MET-driven acquired -resistance.
  * Dose Expansion Phase for participants with evidence of MET-driven acquired -resistance with or without measurable CNS disease.
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Tepotinib — Subjects will receive tepotinib daily in cycles of 21-day duration. Subjects in the Combination Therapy arm will continue to receive their last tolerable dose of tyrosine kinase inhibitor (TKI) together with tepotinib.
  Other Names: Tepmetko

SUMMARY:
This study will look at how effective the study drug (tepotinib) is at stopping the growth and spread of lung cancer with central nervous system metastasis. In some patients, who have developed resistance to their tyrosine kinase inhibitors (TKIs), this study will look at how effective tepotinib is in combination with TKIs. This study will also measure a number of other things including safety of the study drug and the side effects, how body processes the study drug, or how the study drug affects your quality of life.

DETAILED DESCRIPTION:
Phase I - Two arms (Monotherapy and Combination therapy) with primary endpoints of Dose Limiting Toxicity Phase II - Two arms Monotherapy Cohort: Primary endpoint is Intracranial Objective Response Rate Combination Cohort: Primary endpoint is overall and extracranial Objective Response Rate among patients treated with the combination of tepotinib and concurrent TKI.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet ALL of the following criteria are eligible

1. Arm 1 (Monotherapy) Participant has histologic or cytologic confirmation of metastatic MET-driven NSCLC which will be defined by presence of one of the following:

   1. MET Exon 14 skipping mutation as determined by CLIA certified NGS assay. This can be ascertained either by ctDNA based assay or through local testing of tissue samples.
   2. MET amplifications (defined as MET/CEP7 ≥ 4 using FISH)
   3. MET fusions as determined by CLIA certified NGS assay. This can be ascertained either by ctDNA based assay or through local testing for tissue samples.
   4. Other MET driven cases may be considered after consultation and approval by the principal investigator (PI).

   Arm 2 (Combination) Participant has histologic or cytologic confirmation of metastatic NSCLC with documented other driver (eg EGFR or ALK alterations) in which there is evidence of MET-driven acquired resistance (including any of the MET mechanisms noted for dose escalation/CNS expansion monotherapyarms, however due to the potential sub-clonal nature of acquired resistance MET/CEP7 ≥3 or equivalent will explicitly be permitted, or other potential cases with plausible biological evidence after consultation and approval by PI).
2. The participant is able to understand and voluntarily sign a written informed consent and is willing and able to comply with the protocol requirements.
3. Participant is a male or female and at least 18 years of age.
4. Participant has at least 1 measurable lesion by RECIST v1.1 criteria using computed tomography (CT) scan or magnetic resonance image (MRI). Evaluable disease alone will be permitted in the dose escalation cohort. In the CNS efficacy cohort at least one measurable lesion must be intracranial. CNS measurability is defined as below. Measurable CNS lesions ≥10mm in any cohort must be captured as overall and intracranial RECIST target lesions. CNS lesions 5-9mm may be included in intra-cranial data set alone.
5. Participant has an Eastern Cooperative Oncology Group (ECOG) score of 0-2 or Karnofsky score of ≥ 60.
6. Participant has a life expectancy of greater than 12 weeks.
7. Participant is able to ingest oral medications.
8. Participant has received the final dose of any of the following treatments/procedures with the specified minimum intervals before first dose of study drug (unless in the opinion of Investigator and Medical Monitor, the medication will not interfere with study or compromise participant safety).

   Chemotherapy 28 days Antibody drug conjugate (ADC)* 28 days Immune checkpoint inhibitors (ICI) 28 days Stereotactic radiotherapy (SRS) 14 days Tyrosine kinase inhibitor (TKI) † 7 days

   *Prior non-CNS penetrant MET therapy (crizotinib or antibodies directed to MET) is permitted in Arm 1(both dose escalation and CNS Efficacy Evaluation cohort.

   † For patients in Arm 2 (tepotinib for acquired MET resistance), patients will be allowed to remain on their prior TKI without need for a washout therapy. No prior MET therapy within 1 year prior to study start will be allowed for patients being considered forArm 2.
9. Participant has adequate organ function as determined by following laboratory values.

Absolute neutrophil count (ANC)* ≥ 1,500/mm3 (≥ 1.5 x 109/L) Platelets† ≥ 75,000/mm3 (≥ 50 x 109/L) Hemoglobin† ≥ 9 g/dL Serum creatinine ≤ 2 x upper limit normal (ULN) Liver transaminases (ALT/AST) ≤ 3 x ULN

* 5 x ULN, if liver metastases are present on screening Bilirubin ≤ 1.5 x ULN
* 3.0 x ULN, if patient has Gilbert's disease Amylase and lipase ≤ 1.5 x ULN

  * Participants cannot be receiving growth factor support using granulocyte-stimulating colony factor (G-CSF) during the screening visit.

    †Participants cannot receive transfusion support up to one week prior to the screening period.

    10. Participant must meet following radiographic conditions prior to enrollment (CNS expansion cohort)

    a. Measurable, untreated brain metastases (≥ 5mm) will be considered target lesions provided: i. Patient is asymptomatic ii. Patient is on less than 20 mg prednisolone equivalents daily prior to enrolling on study b. Measurable, treated brain metastases (≥ 10mm) growing after whole-brain radiotherapy (WBRT) or resection are allowed as target lesions, but lesions growing after stereotactic radiosurgery (SRS) are allowed as target lesions only if radiation necrosis or pseudoprogression is ruled out.

    c. Leptomeningeal disease (confirmed through either MRI or CSF sampling) is permitted provided this is not the only site of disease. If leptomeningeal disease is present, it will not count as measurable disease.

    11. Female participant of childbearing potential (defined as a sexually mature woman who has not undergone a hysterectomy [surgical removal of the uterus] or bilateral oophorectomy [surgical removal of both ovaries], or if ≥ 45 years old, has not been naturally postmenopausal for at least 24 consecutive months [ie, has had menses at any time during the preceding 24 consecutive months]) must:

    a. Have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.

    b. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) or agree to use and be able to comply with 2 effective methods of contraception without interruption 28 days prior to starting investigational product, during the study therapy (including dose interruptions), and for 120 days after discontinuation (or longer if required by local requirements) of study therapy. The 2 methods of contraception can either be 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy.

    12. Male participant must practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for at least 3 months following investigational product discontinuation (or longer if required by local requirements), even if he has undergone a successful vasectomy.
  * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Note: Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

Participants who meet ANY of the following criteria are not eligible for entry to the study

1. Participant has received an investigational drug within a 28-day period (or within 5 half-lives, whichever is shorter) before the first dose of study drug or is currently participating in another interventional clinical trial, unless in the opinion of the Investigator and Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety.
2. Participants with isolated leptomeningeal disease are not eligible. Patients with symptomatic brain metastases may be potentially eligible provided that all the following criteria are met: 1) they are not on prednisolone 20mg equivalents daily prior to enrolling in the study and 2) anticonvulsants will be permitted provided the patient has been on a stable dose for a period of 2 weeks prior to the first dose of study drug.
3. Participant has clinical evidence or history of ongoing significant bowel obstruction limiting oral intake, active uncontrolled malabsorption syndromes, or any other gastrointestinal disorder or defect that would interfere with absorption, distribution, metabolism, or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity.
4. Participant has New York Association Class III or IV heart failure.
5. Participant has symptomatic acute coronary syndrome, unstable angina, or active ischemia requiring coronary artery stenting, angioplasty, or bypass grafting within 12 weeks prior to starting investigational drug.
6. Participant has evidence of current, uncontrolled, clinically significant, unstable arrhythmias. Participants receiving active anti-arrhythmic therapy are not eligible with the following exceptions:

   1. Participants with atrial fibrillation medically controlled for greater than 1 month prior to Study Day 1.
   2. Participants who have medical pacemakers for control of arrhythmias.
7. Participant has medically uncontrolled hypertension (defined as > 160 mmHg systolic blood pressure (SBP) and > 100 mmHg diastolic blood pressure (DBP).
8. Participant has active/chronic, uncontrolled pancreatitis with serum amylase / lipase ≥ 1.5 ULN.
9. Participant has untreated known HIV/AIDS. Patients with treated and stable HIV (defined as CD4 count >200 cells/mm3 and undetectable HIV viral load) with active, chronic, known outpatient follow up with an HIV specialist will be eligible.
10. Participant has active/chronic, known, untreated, hepatitis B or C infection.
11. Participant has a concurrent and uncontrolled medical illness which would preclude study conduct and assessment, including, but not limited to the following medical conditions: an active infection requiring systemic therapy, bleeding disorder, diabetes mellitus, pulmonary diseases, or alcoholic liver disease.
12. Participant is a pregnant or lactating woman.
13. Participant has a history of severe allergic reactions to any of the study intervention components.
14. Participant has a medical or psychiatric condition, which might compromise their ability to give written informed consent or to comply with the study protocol visits and procedures.
15. Participant has significant reversible toxicities from prior cancer therapy that have not recovered to Grade 1 or baseline (higher grades of alopecia and neuropathy up to Grade 2 will be permitted).
16. Participant has preexisting clinically significant (in the opinion of the investigator) interstitial lung disease or pneumonitis requiring steroid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
ARM 1 (Monotherapy) Dose Limiting Toxicity (DLT) | 1 year
  Dose Escalation Phase: DLT: This is defined as any ≥ to Grade 3 study drug-related toxicity (CTCAE v5.0) occurring within the first cycle of dosing at a given dose level without resolution within 7 days of holding study drug and appropriate supportive care.
Arm 1 (Monotherapy) Intracranial Objective Response Rate (ORR) | 6 years
  Dose Expansion Phase: Intracranial ORR (RECIST 1.1)
Arm 2 (Combination Therapy) Dose Limiting Toxicity (DLT) | 1 year
  Dose Escalation Phase: DLT: This is defined as any ≥ to Grade 3 study drug-related toxicity (CTCAE v5.0) occurring within the first cycle of dosing at a given dose level without resolution within 7 days of holding study drug and appropriate supportive care.
Arm 2 (Combination Therapy) Overall and Extracranial Objective Response Rate | 6 years
  Dose Expansion Phase: Overall and extracranial ORR among patients treated with the combination of tepotinib and concurrent TKI.

SECONDARY OUTCOMES:
ARM 1 (Monotherapy) Blood PK Parameters | 1 year
  Dose escalation phase: Tepotinib blood PK parameters including, but not limited to: Cmax, Tmax, AUC0-t, AUCinf, t1/2, and accumulation ratio.
ARM 1 (Monotherapy) CSF PK Parameters | 1 year
  Dose escalation phase: Tepotinib CSF PK parameters including estimated C8h, C8hrCSF:Cmaxplasma ratio
Arm 1 (Monotherapy) Graded drug-related AEs | 1 year
  Dose escalation phase: To evaluate the frequency of adverse events (AEs) with tepotinib in this patient population.
Arm 1 (Monotherapy) Overall, intracranial and extracranial ORR, PFS, DOR and DCR | 6 years
  Dose expansion phase: Overall, intracranial and extracranial ORR, PFS, DOR and DCR
Arm 1 (Monotherapy) Graded drug-related AEs in CNS efficacy evaluation cohort | 6 years
  Dose expansion phase: Graded drug-related AEs in CNS efficacy evaluation cohort
Arm 2 (Combination) Tepotinib Blood PK Parameters | 1 year
  Dose escalation phase: Tepotinib blood PK parameters including, but not limited to: Cmax, Tmax, AUC0-t, AUCinf, t1/2, and accumulation ratio.
Arm 2 (Combination) Graded drug-related AEs | 1 year
  Dose escalation phase: To evaluate the frequency and severity of AEs with tepotinib in combination with concurrent TKI in patients with MET-driven resistance.
Arm 2 (Combination) Overall, intracranial, and extracranial ORR, PFS, DOR and DCR | 6 years
  Dose Expansion Phase: To evaluate the overall and extracranial ORR, PFS, DOR and DCR among patients treated with the combination of tepotinib and concurrent TKI.
Arm 2 (Combination) Graded drug-related AEs in combination efficacy evaluation cohort | 6 years
  Dose Expansion Phase: To evaluate the frequency and severity of AEs with tepotinib in combination with concurrent TKI in patients with MET-driven resistance.

OTHER OUTCOMES:
Resistance to MET inhibition | 6 years
  Resistance mutations and other mechanisms identified at time of progression on tepotinib.
Overall survival | 6 years
  To estimate the overall survival (OS) among patients treated in each of the cohorts.
Quality of Life Score | 6 years
  Quality of Life score among patients treated in each of the cohorts using the EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: David R Camidge, MD, PhD, Principal Investigator — University of Colorado, Denver; Tejas Patil, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Tyler LC, Le AT, Chen N, Nijmeh H, Bao L, Wilson TR, Chen D, Simmons B, Turner KM, Perusse D, Kasibhatla S, Christiansen J, Dudek AZ, Doebele RC. MET gene amplification is a mechanism of resistance to entrectinib in ROS1+ NSCLC. Thorac Cancer. 2022 Nov;13(21):3032-3041. doi: 10.1111/1759-7714.14656. Epub 2022 Sep 13. PMID 36101520